CLINICAL TRIAL: NCT03773536
Title: Efficacy and Safety of Artesunate + Amodiaquine Combined With a Single Low Dose of Primaquine (0.25 mg/kg) for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Zanzibar
Brief Title: Efficacy and Safety of Artesunate + Amodiaquine With SLD of Primaquine for Treatment of Falciparum Malaria in Zanzibar
Acronym: AcoV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Professor Anders Björkman (Other)
Collaborators: Ministry of Health and Social Welfare, Zanzibar (Other Government); Zanzibar Malaria Elimination Programme (Other Government); Uppsala University (Other)
Responsible Party: Sponsor-Investigator, Professor Anders Björkman, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aco V
Record Dates: First submitted 2018-12-03; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Artesunate-amodiaquine; Single Low Dose Primaquine; Zanzibar
MeSH Terms: conditions — Malaria, Falciparum | interventions — Single Person; Primaquine

STUDY DESIGN:
Intervention Model Description: A one-armed prospective antimalarial drug efficacy trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASAQ + SLD Primaquine (Experimental): Artesunate + amodiaquine (WHO prequalified Artesunate/Amodiaquine Winthrop®) was administered orally as a fixed dose combination, at a dose of approximately artesunate 4 mg/kg + amodiaquine 10mg/kg once daily for 3 consecutive days. Primaquine was administered orally, as a single dose (0.25 mg/kg) together with the first artesunate + amodiaquine dose. All doses of medicine were administered under direct supervision. Any patient who vomited within a 30 minute observation period was re-treated with the same dose of medicine and observed for an additional 30 minutes. If the patient vomited again after the second study drug administration, he/she was withdrawn and offered rescue therapy (Artesunate IV).
  Interventions: Drug: Artesunate-amodiaquine given with single low dose primaquine

INTERVENTIONS:
Drug: Artesunate-amodiaquine given with single low dose primaquine — Three day treatment with ASAQ with SLD primaquine given with the first dose of ASAQ.

SUMMARY:
The general objective of this study is to assess the therapeutic efficacy and safety of artesunate + amodiaquine combined with a single low dose of primaquine (0.25 mg/kg) for the treatment of uncomplicated P. falciparum malaria patients in Zanzibar.

The specific objectives are:

* To determine the clinical and parasitological efficacy of artesunate + amodiaquine and primaquine in the treatment of uncomplicated Plasmodium falciparum infection.
* To differentiate recurrent infections during follow-up, i.e. recrudescence from new infections, by polymerase chain reaction (PCR).
* To evaluate the incidence of adverse events, particularly with regards to potential hematological adverse events of primaquine.
* To determine the polymorphism of molecular markers associated with artesunate + amodiaquine tolerance/resistance.
* To formulate recommendations, which will enable the Zanzibar Ministry of Health to make informed decisions about whether the current national antimalarial treatment guidelines should be updated or not.
* To determine efficacy rate of the first line treatment compared to the first efficacy trial thirteen years ago.

DETAILED DESCRIPTION:
The aim of this study is to provide policymakers with updated efficacy and safety data of artesunate + amodiaquine in combination with a single low dose of primaquine (0.25 mg/kg) and data on genetic markers of tolerance/resistance to artemisinin based combination therapies (ACTs), proposed as an early warning system for development and spread of antimalarial drug resistance, in Zanzibar. The study protocol is based on the new WHO guidelines for surveillance of antimalarial drug efficacy (WHO 2014).

This surveillance study was designed as a one-arm prospective evaluation of the clinical and parasitological responses to directly observed treatment for uncomplicated malaria. Participants were recruited from febrile patients, i.e. documented axillary temperature ≥37.5 °C or history of fever during the past 48 hours, of 3 months and older, presenting at primary health care facilities in Zanzibar, with microscopy confirmed uncomplicated P. falciparum infection. Enrolled patients received directly observed treatment with artesunate + amodiaquine once daily for 3 consecutive days according to the national malaria treatment guidelines. A single low dose of primaquine (0.25 mg/kg) was administered together with the first artesunate + amodiaquine dose. Clinical and parasitological as well as safety parameters were monitored over a 28-day follow-up period. The follow-up consisted of a fixed schedule of check-up visits and corresponding clinical and laboratory examinations. On the basis of the results of these assessments, the patients were classified as having therapeutic failure (early or late) or an adequate response. Blood samples from patients experiencing therapeutic failure during the follow-up period were used to estimate the efficacy of the study drugs based on PCR analysis to distinguish between recrudescence (treatment failures) and reinfection (new infections).

A standard physical examination was performed at baseline (day 0 before drug administration) and on days 1, 2, 3, 7, 14, 21, and 28 ,or any other day if the patient returned spontaneously and parasitological reassessment was required. This examination included measuring axillary temperature, with a thermometer that has a precision of 0.1 °C, as well as conducting a thick film for asexual and gametocyte counts and species identification. Haemoglobin was assessed systematically on all participants on days 0, 3, 7, 14 and 28 using Hemocue, and at any time in case of clinical suspicion of anaemia, i.e. pallor, according to standard case management of malaria in Zanzibar.

In order to differentiate a recrudescence (treatment failure/same parasite strain) from a newly acquired infection (reinfection/different parasite strain) among recurrent parasitemias found during follow-up, a genotype analysis was to be conducted. This analysis was based on the extensive diversity in the following P. falciparum genes: the merozoite surface protein 1 (msp1) and 2 (msp2), and the glutamine-rich protein (glurp) (WHO 2008). The genotypic profiles of pre- and post-parasite strains were to be compared in a stepwise manner to distinguish recrudescence from reinfection. In order to minimize discomfort to the patient due to repeated finger pricks, two to three drops of blood will be collected on a 3MM (Whatman) filter paper during screening or enrollment and each time blood smears are required according to the protocol from day 7.

The results of this study will be used to assist the Zanzibar Ministry of Health in assessing the current national treatment guidelines for uncomplicated P. falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 months and above;
* P. falciparum infection detected by malaria rapid diagnostic test (mRDT) and confirmed by microscopy;
* Presence of P. falciparum malaria asexual parasitaemia (any level);
* Presence of axillary ≥37.5 °C or history of fever during the past 48 hours
* Ability to swallow oral medication;
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* Informed consent from the patient or from a parent or guardian in the case of children.

Exclusion Criteria:

* Presence of general danger signs in children aged under 5 years or signs of severe falciparum malaria according to the definitions of WHO (Appendix 1);
* Mono-infection with a Plasmodium species other than P. falciparum detected by microscopy;
* Presence of febrile conditions other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. severe malnutrition, cardiac, renal and hepatic diseases, HIV/AIDS);
* Regular medication, which may interfere with the study drugs;
* History of hypersensitivity reactions or contraindications to any of the study medicines; and
* Pregnancy

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
PCR corrected cure rates for assessing efficacy of artesunate + amodiaquine given together with a single low dose primaquine in the treatment of uncomplicated Plasmodium falciparum infection | 42 days
  PCR corrected cure rates were to be assessed by genotype analysis of the following P. falciparum genes: the merozoite surface protein 1 (msp1) and 2 (msp2), and the glutamine-rich protein (glurp) (WHO 2008). The genotypic profiles of pre- and post-parasite strains were to be compared in a stepwise manner to distinguish recrudescence from reinfection.

SECONDARY OUTCOMES:
Safety of artesunate + amodiaquine and primaquine: Incidence of adverse events | 42 days
  Incidence of adverse events, particularly with regards to potential hematological adverse events of primaquine.

OTHER OUTCOMES:
Monitoring molecular markers of drug resistance | 42 days
  Prevalence of genetic polymorphisms associated with artesunate + amodiaquine tolerance/resistance. I.e., prevalence of genetic markers in the P. falciparum chloroquine resistance transporter gene (pfcrt), the multidrug resistance gene 1 (pfmdr1), and in the Kelch 13 propeller region.

CONTACTS AND LOCATIONS:
Overall Officials: Mwinyi I Msellem, Principal Investigator — Mnazi mmoja hospital, Zanzibar Ministry of Health; Abduallah S Ali, Study Director — Zanzibar Malaria Elimination Programme; Andreas Martensson, Study Chair — Uppsala University
Locations (1):
- Micheweni, Bububu Jesheni, and Uzini, Zanzibar, Tanzania

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03773536/Prot_SAP_ICF_000.pdf